CLINICAL TRIAL: NCT06081452
Title: Public Survey on Breath Testing for Health and Disease
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 6634264
Record Dates: First submitted 2023-10-06; First posted 2023-10-13 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Disease; Health Behavior; Health Attitude; Health-Related Behavior; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Neoplasms; Disease; Health Behavior; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Public: General public to be approached to answer this survey via GPs, charities and exhibitions such as Great Exhibition Road Festival.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Members of the public will be asked to complete a survey that collects information on individuals perception of health and disease and their views on breath testing.

SUMMARY:
A brief survey for the public to determine interest in health surveillance and disease detection

DETAILED DESCRIPTION:
There are numerous barriers and favourable conditions that affect the acceptability of a screening test for cancer. Such factors have been investigated in the context of some of the current screening programs. Through this survey the investigators want to increase researcher awareness of these factors with the hope that this information will aid policy makers and guide future research.

There has been widening public interest in general health-surveillance in addition to disease detection. Breath testing has the potential to be a one-for-all non-invasive test to detect health domains. Through this survey, the investigators wish to understand public opinions about breath testing for health.

This survey consists of questions aiming to gather views on non-invasive testing for health and disease.

ELIGIBILITY:
Inclusion Criteria:

* Member of the public above the age of 18

Exclusion Criteria:

* Member of the public below the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our aim is to acquire a wide breadth of information from all members of the public, irrespective of the demographics, socioeconomic status and ethnicity. All member of the public, above the age of 18 are welcome to participate
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-17 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Acceptability of breath testing | 6 months
  Proportion of people that find breath testing an acceptable means to determine health or disease

CONTACTS AND LOCATIONS:
Overall Officials: George Hanna, PhD, Study Director — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided